CLINICAL TRIAL: NCT00759876
Title: A Phase 2a Extension Study of PTC124 in Subjects With Nonsense-Mutation-Mediated Duchenne Muscular Dystrophy
Brief Title: Phase 2a Extension Study of Ataluren (PTC124) in Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early because similar study with Ataluren (PTC124-GD-007-DMD; NCT00592553) exhibited lack of efficacy at the high dose (not due to safety concerns).
Sponsor: PTC Therapeutics (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-004e-DMD
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Nonsense mutation; Premature stop codon; DMD; PTC124; Ataluren
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren (Experimental): Participants will receive ataluren 3 times per day with meals at doses of 20 milligrams per kilogram (mg/kg) (breakfast), 20 mg/kg (lunch), and 40 mg/kg (dinner) for up to 89 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with milk. Dosing based on participant body weight
  Other Names: PTC124

SUMMARY:
Duchenne muscular dystrophy (DMD) is a genetic disorder that develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability during childhood and teenage years. A specific type of mutation, called a nonsense (premature stop codon) mutation, is the cause of DMD in approximately 10-15% of boys with the disease. Ataluren is an orally-delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 2a extension trial that will evaluate the long-term safety of ataluren in boys with nonsense mutation DMD, as determined by adverse events and laboratory abnormalities. The study will also assess changes in walking, muscle function, strength, and other important clinical and laboratory measures.

DETAILED DESCRIPTION:
This Phase 2a, multicenter, open-label safety and efficacy study will be performed at 3 sites in the United States. The study will enroll up to 38 participants with nonsense mutation Duchenne muscular dystrophy who participated in a previous Phase 2a study of ataluren (Protocol Number PTC124-GD-004-DMD [NCT00264888]). Participants will receive study drug 3 times per day (at breakfast, lunch, and dinner) for approximately 96 weeks (approximately 2 years). Study assessments will be performed at clinic visits during screening, every 6 weeks for the first 24 weeks, and then every 12 weeks until the end of the study. Additional safety laboratory testing, which may be performed at the investigational site or at an accredited local laboratory or clinic, is required every 3 weeks for the first 24 weeks and then every 6 weeks from Week 24 to Week 48. Participants will have a biceps muscle biopsy before ataluren treatment and again after 24 weeks of ataluren treatment to evaluate changes in muscle dystrophin expression. An evaluation of the effects of ataluren on corticosteroid pharmacokinetics will be performed. Associated with this ataluren clinical trial is a substudy that will use magnetic resonance evaluations to assess changes in the composition of muscles of the legs.

ELIGIBILITY:
Inclusion Criteria:

* Completion of ataluren treatment in the previous Phase 2a study (Protocol PTC124-GD-004-DMD).
* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if <18 years of age).
* Confirmed screening laboratory values within the central laboratory ranges.
* In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during ataluren administration and the 6-week follow up period.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Treatment with systemic aminoglycoside antibiotics within 3 months prior to start of study treatment.
* Treatment with warfarin within 1 month prior to start of study treatment.
* Known hypersensitivity to any of the ingredients or excipients of the study drug (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab-O-Sil® M5P [colloidal silica], and magnesium stearate).
* Exposure to another investigational drug within 2 months prior to start of study treatment.
* History of major surgical procedure within 1 month prior to start of study treatment.
* Ongoing immunosuppressive therapy (other than corticosteroids).
* Ongoing participation in any other clinical trial (except for sub-studies specifically approved by PTC Therapeutics).
* Clinically significant symptoms and signs of congestive heart failure (CHF) (American College of Cardiology/American Heart Association Stage C or Stage D).
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, electrocardiogram findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants only are being studied.
Enrollment: 36 (Actual)
Dates: Start 2008-08-13 (Actual); Primary Completion 2010-05-17 (Actual); Study Completion 2010-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leone Atkinson, Study Director — PTC Therapeutics, Inc.
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- [Background] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- See also: Related Info — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was initiated approximately 2 years after the completion of Study PTC124-GD-004-DMD (Study 004 [NCT00264888]).
Pre-assignment Details: Of the 36 participants, 11 received 20-, 20-, and 40-milligrams/kilograms (mg/kg); 20 received 10-, 10-, and 20-mg/kg; and 5 received 4-, 4-, and 8-mg/kg ataluren dose level in Study 004. The 31 participants receiving corticosteroid treatment at study entry could continue corticosteroid treatment during the study as long as regimen remained stable.
Groups:
- Ataluren: Participants received ataluren 3 times per day with meals at doses of 20 mg/kg (breakfast), 20 mg/kg (lunch), and 40 mg/kg (dinner) for up to 89 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 36
As-Treated Population (All participants who received at least 1 dose of study drug in this study.) | 36
Evaluable Population (Participants in the As-Treated Population with Baseline and on-treatment data in this study.) | 35
Ambulatory Evaluable Population (Participants with the ability to walk ≥75 meters unassisted at screening.) | 24
Completed | 0
Not Completed | 36
Not completed — Sponsor terminated study early | 36

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population).
Arm/Group | Ataluren
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAE: any untoward medical occurrence or undesirable event(s) that begins or worsens following administration of the study drug, whether or not considered related to the treatment by the Investigator. Severity of an adverse event (AE) was classified as: mild (does not interfere with usual function), moderate (interferes with usual function; may require medical intervention), severe (interferes significantly with usual function; likely require medical intervention), life-threatening, and fatal. Drug-related AEs: AEs with a possible or probable relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 89
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 36
Participants
  At least 1 TEAE | 36
  Mild TEAE | 9
  Moderate TEAE | 16
  Severe TEAE | 10
  Life-Threatening TEAE | 1
  Fatal TEAE | 0
  Related TEAE | 28
  Serious TEAE | 6

2. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) as Measured by the 6-minute Walk Test (6MWT)
Description: The 6MWD was assessed in participants who were ambulatory using standardized procedures. Participants were not permitted to use assistive devices during the 6MWD test. Only the results of the participant's best valid test at each visit were included in the analysis. The mean change from baseline in the distance the participant walked is reported.
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable 6MWT data. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ataluren
Number analyzed (Participants) | 23
meters
  Baseline | 367.8 (107.3)
  Change from Baseline at Week 48: number analyzed (Participants) | 22
  Change from Baseline at Week 48 | -80.4 (59.5)
  Change from Baseline at Week 60: number analyzed (Participants) | 19
  Change from Baseline at Week 60 | -101.5 (64.4)

3. Secondary Outcome: Change From Baseline in Proximal Muscle Function as Assessed by Speed During Timed Function Tests
Description: Timed function tests included time to stand from supine position (rise to standing), time to run/walk 10 meters (m), and time to ascend/descend 4 stairs. Timed function tests were assessed in ambulatory participants. A decrease from baseline reflects faster completion of the functional task and, thus, better muscle function. If the time taken to perform a test exceeded 30 seconds or if a participant could not perform the test due to disease progression (PD), a value of 30 seconds was used. Test results were set to missing in the analysis for participants who could not perform the tests for reasons other than PD (for example, bone fracture).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable data for the applicable timed function test. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 24
seconds
  Rise to Standing, Baseline | 13.57 (11.111)
  Rise to Standing, Change from Baseline at Week 48 | 6.49 (8.059)
  Rise to Standing, Change from Baseline at Week 60: number analyzed (Participants) | 21
  Rise to Standing, Change from Baseline at Week 60 | 5.77 (7.790)
  Walk/Run 10 m, Baseline | 7.62 (3.641)
  Walk/Run 10 m, Change from Baseline at Week 48 | 3.15 (5.591)
  Walk/Run 10 m, Change from Baseline at Week 60: number analyzed (Participants) | 21
  Walk/Run 10 m, Change from Baseline at Week 60 | 3.20 (5.930)
  Ascend 4 Stairs, Baseline | 7.16 (7.481)
  Ascend 4 Stairs, Change from Baseline at Week 48 | 4.92 (6.856)
  Ascend 4 Stairs, Change from Baseline at Week 60: number analyzed (Participants) | 21
  Ascend 4 Stairs, Change from Baseline at Week 60 | 6.30 (7.926)
  Descend 4 Stairs, Baseline | 6.42 (7.565)
  Descend 4 Stairs, Change from Baseline at Week 48 | 5.25 (8.839)
  Descend 4 Stairs, Change from Baseline at Week 60: number analyzed (Participants) | 21
  Descend 4 Stairs, Change from Baseline at Week 60 | 4.28 (7.275)

4. Secondary Outcome: Change From Baseline in Standing From Supine Position as Assessed by Method Scores During Timed Function Tests
Description: Timed test evaluations included scoring of method that ambulatory participants used to complete test. Scale for method used for standing from supine position: 1) Unable to stand from supine, even with use of a chair. 2) Assisted Gowers, requires furniture to rise from supine to full upright posture. 3) Full Gowers, rolls over, stands with both hands "climbing up" legs to above knees to achieve full upright posture. 4) Half Gowers, rolls over, stands up with 1 hand support on lower legs. 5) Rolls to side and/or stands with 1 or both hands on floor to start to rise but does not touch legs. 6) Stands without rolling over or using hands. Increases from baseline are indicative of improving ability to perform functional task. If a participant could not perform a timed function test because of PD, a method value of "1" was assigned in analysis. Test results set to missing in analysis for participants who could not perform tests for reasons other than PD (for example, bone fracture).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable method data for standing from supine. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 24
scores on a scale
  Baseline | 3.25 (1.260)
  Change from Baseline at Week 48 | -0.58 (0.929)
  Change from Baseline at Week 60: number analyzed (Participants) | 21
  Change from Baseline at Week 60 | -0.62 (0.921)

5. Secondary Outcome: Change From Baseline in Run/Walk 10-Meters as Assessed by Method Scores During Timed Function Tests
Description: Timed test evaluations included scoring of method that ambulatory participants used to complete test. Scale for method used to run/walk 10-meters: 1) Unable to walk independently. 2) Unable to walk independently but can walk with knee-ankle-foot orthoses (KAFOs) or with support from a person 3) Highly adapted, wide-based lordotic gait, cannot increase walking speed. 4) Moderately adapted gait, can pick up speed but cannot run. 5) Able to pick up speed but runs with a double stance phase (that is, cannot achieve both feet off the ground). 6) Runs and gets both feet off the ground (with no double-stance phase). At the visit, if a participant could not perform a timed function test because of PD, a method value of "1" was assigned in analysis. Test results set to missing in analysis for participants who could not perform tests for reasons other than PD (for example, bone fracture).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable method data for running/walking 10 meters. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 24
scores on a scale
  Baseline | 4.42 (0.974)
  Change from Baseline at Week 48 | -0.25 (1.073)
  Change from Baseline at Week 60: number analyzed (Participants) | 21
  Change from Baseline at Week 60 | -0.57 (1.207)

6. Secondary Outcome: Change From Baseline in Ascending 4 Stairs as Assessed by Method Scores During Timed Function Tests
Description: Timed test evaluations included scoring of method that ambulatory participants used to complete test. Scale for method used to ascend 4 stairs: 1) Unable to climb 4 standard stairs. 2) Climbs 4 standard stairs "marking time" (climbs 1 foot at a time, with both feet on a step before moving to next step), using both arms on 1 or both handrails. 3) Climbs 4 standard stairs "marking time" using 1 arm on 1 handrail. 4) Climbs 4 standard stairs "marking time" not needing handrail. 5) Climbs 4 standard stairs alternating feet, needs handrail for support. 6) Climbs 4 standard stairs alternating feet, not needing handrail support. At the visit, if a participant could not perform a timed function test because of PD, a method value of "1" was assigned in analysis. Test results set to missing in analysis for participants who could not perform tests for reasons other than PD (for example, bone fracture).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable method data for ascending 4 stairs. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 24
scores on a scale
  Baseline | 3.58 (1.717)
  Change from Baseline at Week 48 | -0.46 (1.141)
  Change from Baseline at Week 60: number analyzed (Participants) | 21
  Change from Baseline at Week 60 | -0.48 (1.365)

7. Secondary Outcome: Change From Baseline in Descending 4 Stairs as Assessed by Method Scores During Timed Function Tests
Description: Timed test evaluations included scoring of method that ambulatory participants used to complete test. Scale for method used to descend 4 stairs: 1) Unable to descend 4 standard stairs. 2) Descends 4 standard stairs "marking time" (climbs 1 foot at a time, with both feet on a step before moving to next step), using both arms on 1 or both handrails. 3) Descends 4 standard stairs "marking time", using 1 arm on 1 handrail. 4) Descends 4 standard stairs "marking time", not needing handrail. 5) Descends 4 standard stairs alternating feet in both directions, needs handrail for support. 6) Descends 4 standard stairs alternating feet, not needing handrail support. At the visit, if a participant could not perform a timed function test because of PD, a method value of "1" was assigned in analysis. Test results set to missing in analysis for participants who could not perform tests for reasons other than PD (for example, bone fracture).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable method data for descending 4 stairs. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 24
scores on a scale
  Baseline | 3.63 (1.740)
  Change from Baseline at Week 48 | -0.04 (1.160)
  Change from Baseline at Week 60: number analyzed (Participants) | 21
  Change from Baseline at Week 60 | -0.10 (0.889)

8. Secondary Outcome: Change From Baseline in Force Exerted During Knee Flexion and Extension, Elbow Flexion and Extension, Shoulder Abduction, and Hand Grip as Assessed by Myometry
Description: Upper extremity myometry was performed using a hand-held dynamometer following standardized procedures. With this system, evaluators judged the strength of each muscle using an 11-point descriptive scoring system. From the individual muscle-group scores, a total composite score was derived. Bilateral assessments were done, and 3 measurements were recorded from each muscle group on each side, when possible. The best of the 3 replicates was used in the analysis. An increase from Baseline is reflective of increased muscle strength, whereas a decrease from Baseline is reflective of decreased muscle strength. Participants who became unable to perform a myometry test because of disease progression were assigned a value of 0 for each visit at which the participant was no longer able to perform the test. Test results were set to missing in the analysis for participants who could not perform the tests for reasons other than disease progression (for example, bone fracture).
Time Frame: Baseline, Week (Wk) 48 and Wk 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable myometry data.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Ataluren
Number analyzed (Participants) | 35
pounds
  Left (L) Knee Flexion, Baseline | 9.48 (4.395)
  L Knee Flexion, Change from Baseline at Wk 48 | 1.23 (2.715)
  L Knee Flexion, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  L Knee Flexion, Change from Baseline at Wk 60 | 0.64 (3.079)
  Right (R) Knee Flexion, Baseline | 10.15 (5.439)
  R Knee Flexion, Change from Baseline at Wk 48 | 0.81 (2.254)
  R Knee Flexion, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  R Knee Flexion, Change from Baseline at Wk 60 | -0.05 (2.240)
  L Knee Extension, Baseline | 8.63 (5.124)
  L Knee Extension, Change from Baseline at Wk 48 | -1.07 (1.842)
  L Knee Extension, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  L Knee Extension, Change from Baseline at Wk 60 | -1.00 (1.567)
  R Knee Extension, Baseline | 9.10 (6.109)
  R Knee Extension, Change from Baseline at Wk 48 | -1.33 (2.021)
  R Knee Extension, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  R Knee Extension, Change from Baseline at Wk 60 | -1.65 (2.204)
  L Elbow Flexion, Baseline | 5.70 (3.611)
  L Elbow Flexion, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  L Elbow Flexion, Change from Baseline at Wk 48 | -0.15 (0.998)
  L Elbow Flexion, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  L Elbow Flexion, Change from Baseline at Wk 60 | -0.51 (1.121)
  R Elbow Flexion, Baseline | 5.85 (3.758)
  R Elbow Flexion, Change from Baseline at Wk 48: number analyzed (Participants) | 33
  R Elbow Flexion, Change from Baseline at Wk 48 | -0.28 (1.050)
  R Elbow Flexion, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  R Elbow Flexion, Change from Baseline at Wk 60 | -0.55 (1.061)
  L Elbow Extension, Baseline | 4.55 (2.322)
  L Elbow Extension, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  L Elbow Extension, Change from Baseline at Wk 48 | -0.10 (0.993)
  L Elbow Extension, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  L Elbow Extension, Change from Baseline at Wk 60 | -0.32 (0.818)
  R Elbow Extension, Baseline | 4.89 (2.680)
  R Elbow Extension, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  R Elbow Extension, Change from Baseline at Wk 48 | -0.10 (1.600)
  R Elbow Extension, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  R Elbow Extension, Change from Baseline at Wk 60 | -0.60 (1.352)
  L Shoulder Abduction, Baseline | 4.29 (2.783)
  L Shoulder Abduction Change from Baseline at Wk 48: number analyzed (Participants) | 27
  L Shoulder Abduction Change from Baseline at Wk 48 | -0.90 (0.906)
  L Shoulder Abduction Change from Baseline at Wk 60: number analyzed (Participants) | 23
  L Shoulder Abduction Change from Baseline at Wk 60 | -1.10 (1.632)
  R Shoulder Abduction, Baseline: number analyzed (Participants) | 31
  R Shoulder Abduction, Baseline | 4.39 (2.666)
  R Shoulder Abduction Change from Baseline at Wk 48: number analyzed (Participants) | 26
  R Shoulder Abduction Change from Baseline at Wk 48 | -1.02 (1.369)
  R Shoulder Abduction Change from Baseline at Wk 60: number analyzed (Participants) | 21
  R Shoulder Abduction Change from Baseline at Wk 60 | -1.23 (1.888)
  L Hand Grip, Baseline | 15.19 (5.881)
  L Hand Grip, Change from Baseline at Wk 48 | 0.30 (3.353)
  L Hand Grip, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  L Hand Grip, Change from Baseline at Wk 60 | 1.04 (4.811)
  R Hand Grip, Baseline | 17.17 (7.266)
  R Hand Grip, Change from Baseline at Wk 48 | -0.79 (3.628)
  R Hand Grip, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  R Hand Grip, Change from Baseline at Wk 60 | -0.61 (3.010)

9. Secondary Outcome: Change in Resting, Active, and Recovery Heart Rate as Assessed by Heart Rate Monitoring With the Polar RS400
Description: Heart rate was measured with a Polar RS400 heart rate monitor, which consists of a transmitter strap worn around the chest and a wristwatch receiver. The monitor produces a digital text file with 1 value per minute that represents the mean heart rate for that minute. Mean heart rate values were collected before, during, and after the 6MWT. The participant rested for 5 minutes in a sitting position before the 6MWT, and the mean heart rate for the last minute of this rest period was obtained and documented as the resting heart rate. During the 6MWT, the mean heart rate was collected and documented as the active heart rate. After completing the 6MWT and resting for 3 minutes, the mean heart rate for 1 minute was obtained and documented as the recovery heart rate.
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable heart rate data. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: beeps per minute
Arm/Group | Ataluren
Number analyzed (Participants) | 24
beeps per minute
  Resting Heart Rate, Baseline | 106.46 (11.163)
  Resting Heart Rate, Change from Baseline at Wk 48: number analyzed (Participants) | 23
  Resting Heart Rate, Change from Baseline at Wk 48 | 8.30 (12.382)
  Resting Heart Rate, Change from Baseline at Wk 60: number analyzed (Participants) | 19
  Resting Heart Rate, Change from Baseline at Wk 60 | 5.16 (11.197)
  Active Heart Rate, Baseline | 152.17 (13.457)
  Active Heart Rate, Change from Baseline at Wk 48: number analyzed (Participants) | 22
  Active Heart Rate, Change from Baseline at Wk 48 | 3.86 (12.365)
  Active Heart Rate, Change from Baseline at Wk 60: number analyzed (Participants) | 19
  Active Heart Rate, Change from Baseline at Wk 60 | -2.84 (17.238)
  Recovery Heart Rate, Baseline | 113.13 (12.664)
  Recovery Heart Rate, Change from Baseline at Wk 48: number analyzed (Participants) | 22
  Recovery Heart Rate, Change from Baseline at Wk 48 | 4.64 (9.079)
  Recovery Heart Rate, Change from Baseline at Wk 60: number analyzed (Participants) | 19
  Recovery Heart Rate, Change from Baseline at Wk 60 | 1.68 (15.688)

10. Secondary Outcome: Change From Baseline in Verbal Memory and Attention as Assessed by the Digit Span Task
Description: The digit span task is a 2-part (forward and backward) test in which a series of digits (3 to 9) were presented to participant in an auditory format only. For forward condition, the participant was to repeat digits back in the order they were presented. For backward condition, the participant was to reverse the order of presentation. Maximum score for each part (digit forward and digit backward) of task is 14; participants received a score of 2 points if they passed both trials, score of 1 point if they passed only 1 trial, and score of 0 points if they failed both trials. A raw score of total number of correct forward and backward responses was age-normalized by subtracting corresponding mean and dividing by corresponding standard deviation of a reference population for that age. For each forward and backward result, the resulting Z score was transformed into percentile rank of normal distribution. Change from Baseline in number of digits recalled forward and backward is reported.
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable verbal memory and attention data.
Measure: Mean (Standard Deviation); unit: digits recalled
Arm/Group | Ataluren
Number analyzed (Participants) | 35
digits recalled
  Recalled Forward, Baseline | 3.66 (2.378)
  Recalled Forward, Change from Baseline at Wk 48 | 0.14 (1.353)
  Recalled Forward, Change from Baseline at Wk 60: number analyzed (Participants) | 28
  Recalled Forward, Change from Baseline at Wk 60 | 0.04 (1.453)
  Recalled Backward, Baseline: number analyzed (Participants) | 34
  Recalled Backward, Baseline | 3.15 (2.524)
  Recalled Backward, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Recalled Backward, Change from Baseline at Wk 48 | 0.74 (1.442)
  Recalled Backward, Change from Baseline at Wk 60: number analyzed (Participants) | 34
  Recalled Backward, Change from Baseline at Wk 60 | 0.74 (1.442)

11. Secondary Outcome: Change From Baseline in Participant-Reported Health-Related Quality of Life (HRQL) as Measured by the Pediatric Quality of Life Inventory (PedsQL) Inventory
Description: The PedsQL Generic Core Scales comprises 23 questions, which are grouped into 4 scales (physical functioning, emotional functioning, social functioning, and school functioning); the fatigue-specific module included an additional 18 questions. The appropriate age-specific version was completed. On PedsQL Generic Core Scales, items were reversed scored and linearly transformed to a 0 to 100 scale so that higher scores indicate a better HRQL (0=100, 1=75, 2=50, 3=25, and 4=0). Mean is the sum of the items over the number of items that were answered (which accounts for missing data) to create scale scores. If >50% of the items in a scale were missing, the scale score was not computed. Mean Total Scale Score is the sum of all of the items over the number of items that were answered on all scales.
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable participant-reported PedsQL data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 35
scores on a scale
  Physical Functioning, Baseline: number analyzed (Participants) | 34
  Physical Functioning, Baseline | 45.13 (21.114)
  Physical Functioning Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Physical Functioning Change from Baseline at Wk 48 | 3.16 (20.180)
  Physical Functioning Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Physical Functioning Change from Baseline at Wk 60 | 6.25 (23.545)
  Emotional Functioning, Baseline: number analyzed (Participants) | 34
  Emotional Functioning, Baseline | 65.29 (16.141)
  Emotional Function, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Emotional Function, Change from Baseline at Wk 48 | 8.24 (18.294)
  Emotional Function, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Emotional Function, Change from Baseline at Wk 60 | 12.22 (17.614)
  Social Functioning, Baseline: number analyzed (Participants) | 34
  Social Functioning, Baseline | 61.80 (16.914)
  Social Functioning, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Social Functioning, Change from Baseline at Wk 48 | 4.82 (19.463)
  Social Functioning, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Social Functioning, Change from Baseline at Wk 60 | 3.75 (15.861)
  School Functioning, Baseline: number analyzed (Participants) | 34
  School Functioning, Baseline | 70.29 (16.466)
  School Functioning, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  School Functioning, Change from Baseline at Wk 48 | 1.76 (17.917)
  School Functioning, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  School Functioning, Change from Baseline at Wk 60 | 3.29 (16.273)
  Fatigue Scale Score, Baseline: number analyzed (Participants) | 34
  Fatigue Scale Score, Baseline | 74.28 (14.917)
  Fatigue Scale Score, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Fatigue Scale Score, Change from Baseline at Wk 48 | 5.08 (12.661)
  Fatigue Scale Score, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Fatigue Scale Score, Change from Baseline at Wk 60 | 4.39 (11.777)
  Total Score, Baseline: number analyzed (Participants) | 34
  Total Score, Baseline | 58.59 (12.793)
  Total Score, Change from Baseline at Wk 48: number analyzed (Participants) | 34
  Total Score, Change from Baseline at Wk 48 | 4.28 (13.406)
  Total Score, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Total Score, Change from Baseline at Wk 60 | 6.42 (10.887)

12. Secondary Outcome: Change From Baseline in Parent- or Caregiver-Reported HRQL as Measured by the PedsQL Inventory
Description: The PedsQL Generic Core Scales comprises 23 questions, which are grouped into 4 scales (physical functioning, emotional functioning, social functioning, and school functioning); the fatigue-specific module included an additional 18 questions. The appropriate age-specific version was completed. On PedsQL Generic Core Scales, items were reversed scored and linearly transformed to a 0 to 100 scale so that higher scores indicate a better HRQL (0=100, 1=75, 2=50, 3=25, and 4=0). Mean is the sum of the items over the number of items that were answered (which accounts for missing data) to create scale scores. If >50% of the items in a scale were missing, the scale score was not computed. Mean Fatigue Scale Score is the sum of the items over the number of items that were answered in the Emotional, Social, and School Functioning Scales. Mean Total Scale Score is the sum of all of the items over the number of items that were answered on all scales.
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable parent- or caregiver-reported PedsQL data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 35
scores on a scale
  Physical Functioning, Baseline: number analyzed (Participants) | 34
  Physical Functioning, Baseline | 48.07 (21.111)
  Physical Functioning Change from Baseline at Wk 48: number analyzed (Participants) | 33
  Physical Functioning Change from Baseline at Wk 48 | 2.31 (20.284)
  Physical Functioning Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Physical Functioning Change from Baseline at Wk 60 | 1.85 (19.366)
  Emotional Functioning, Baseline: number analyzed (Participants) | 34
  Emotional Functioning, Baseline | 69.45 (17.465)
  Emotional Function, Change from Baseline at Wk 48: number analyzed (Participants) | 33
  Emotional Function, Change from Baseline at Wk 48 | 5.27 (19.595)
  Emotional Function, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Emotional Function, Change from Baseline at Wk 60 | 3.29 (20.021)
  Social Functioning, Baseline: number analyzed (Participants) | 34
  Social Functioning, Baseline | 57.95 (19.397)
  Social Functioning, Change from Baseline at Wk 48: number analyzed (Participants) | 33
  Social Functioning, Change from Baseline at Wk 48 | 9.38 (16.956)
  Social Functioning, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Social Functioning, Change from Baseline at Wk 60 | 6.16 (17.599)
  School Functioning, Baseline: number analyzed (Participants) | 34
  School Functioning, Baseline | 67.61 (14.944)
  School Functioning, Change from Baseline at Wk 48: number analyzed (Participants) | 32
  School Functioning, Change from Baseline at Wk 48 | 5.66 (15.824)
  School Functioning, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  School Functioning, Change from Baseline at Wk 60 | -0.37 (10.651)
  Fatigue Scale Score, Baseline: number analyzed (Participants) | 34
  Fatigue Scale Score, Baseline | 72.25 (13.777)
  Fatigue Scale Score, Change from Baseline at Wk 48: number analyzed (Participants) | 33
  Fatigue Scale Score, Change from Baseline at Wk 48 | 0.77 (9.703)
  Fatigue Scale Score, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Fatigue Scale Score, Change from Baseline at Wk 60 | -0.40 (9.269)
  Total Score, Baseline: number analyzed (Participants) | 34
  Total Score, Baseline | 59.08 (13.348)
  Total Score, Change from Baseline at Wk 48: number analyzed (Participants) | 33
  Total Score, Change from Baseline at Wk 48 | 5.24 (11.409)
  Total Score, Change from Baseline at Wk 60: number analyzed (Participants) | 27
  Total Score, Change from Baseline at Wk 60 | 2.68 (12.261)

13. Secondary Outcome: Change From Baseline in Serum Creatine Kinase (CK) Levels
Description: Serum CK concentrations (as measured by the central laboratory) were quantified from the blood samples that were collected as part of the safety laboratory evaluations. The normal range for CK is 18 to 363 units/liter (U/L).
Time Frame: Baseline, Week 48 and Week 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable CK data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ataluren
Number analyzed (Participants) | 35
U/L
  Baseline | 5988.31 (3967.714)
  Change from Baseline at Week 48: number analyzed (Participants) | 34
  Change from Baseline at Week 48 | 84.06 (2641.422)
  Change from Baseline at Week 60: number analyzed (Participants) | 28
  Change from Baseline at Week 60 | -549.57 (3261.151)

14. Secondary Outcome: Change From Baseline in Dystrophin Expression on Biceps Muscle Biopsy as Measured by Immunofluorescence Staining of the Sarcolemmal Membrane With an Antibody to the C-Terminal Portion of the Dystrophin Protein
Description: The biceps muscle was biopsied from 1 arm for confirmation of the absence or low levels of dystrophin prior to treatment initiation and from the other arm to assess for production of dystrophin post-treatment. Muscle tissue sections were processed and immunostained to detect muscle membrane-localized dystrophin. An increase in value indicates dystrophin production.
Time Frame: Baseline, Week 24
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population) and had evaluable dystrophin expression data.
Measure: Mean (Standard Deviation); unit: dystrophin positive fibers
Arm/Group | Ataluren
Number analyzed (Participants) | 36
dystrophin positive fibers
  Baseline | 16.828 (8.4285)
  Change from Baseline: number analyzed (Participants) | 35
  Change from Baseline | -1.880 (5.1337)

15. Secondary Outcome: Study Drug Compliance
Description: Study drug compliance was assessed by the participant daily diary and quantification of used and unused study drug. Compliance was assessed in terms of the amount of drug actually taken relative to the amount that was prescribed. Physician-prescribed dose reductions and interruptions were factored into the calculations. "Not recorded" applies only to the days on which all dosing information was missing or for missing days. Invalid entries in the participant daily diary were assigned values of 0.0 for percentage of doses taken and 99.0 for percentage of doses not recorded.
Time Frame: Baseline up to Week 89
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population).
Measure: Median (Full Range); unit: percentage of doses of study drug
Arm/Group | Ataluren
Number analyzed (Participants) | 36
percentage of doses of study drug
  Percentage of Doses Taken as Planned | 84.7 [0 to 99.2]
  Percentage of Doses Missed | 1.1 [0 to 13.2]
  Percentage of Doses Changed | 0.3 [0 to 22.2]
  Percentage of Doses Not Recorded | 10.2 [0 to 99.0]

16. Secondary Outcome: Pharmacokinetics: Ataluren Plasma Exposure in All Participants
Description: Blood for ataluren concentrations over a 24-hour period was to be collected on Day 2 of Week 1 and Day 2 of Week 6. Analysis of the blood samples was to be conducted using a validated high-performance liquid chromatography with tandem mass spectrometry (HPLC-MS/MS) method with a lower limit of quantitation (LLOQ) of 0.5 micrograms/milliliters (μg/mL). Plasma concentrations below qualification (BQ) is treated as 0 in the summary calculation.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, and 4 hours post-morning dose and 0 (pre-dose) and 2 hours post-midday dose on Day 2 of Week 1 and Day 2 of Week 6
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population) and had evaluable plasma data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 36
μg/mL
  Pre-Morning Dose, Week 1: number analyzed (Participants) | 35
  Pre-Morning Dose, Week 1 | 0 (0)
  30 minutes Post-Morning Dose, Week 1: number analyzed (Participants) | 33
  30 minutes Post-Morning Dose, Week 1 | 14.59 (10.404)
  1 hour Post-Morning Dose, Week 1: number analyzed (Participants) | 34
  1 hour Post-Morning Dose, Week 1 | 16.24 (10.251)
  2 hours Post-Morning Dose, Week 1: number analyzed (Participants) | 34
  2 hours Post-Morning Dose, Week 1 | 23.71 (12.895)
  3 hours Post-Dose, Week 1: number analyzed (Participants) | 34
  3 hours Post-Dose, Week 1 | 28.96 (15.306)
  4 hours Post-Morning Dose, Week 1: number analyzed (Participants) | 34
  4 hours Post-Morning Dose, Week 1 | 29.44 (14.854)
  Pre-Midday Dose, Week 1: number analyzed (Participants) | 34
  Pre-Midday Dose, Week 1 | 20.43 (15.256)
  2 hours Post-Midday Dose, Week 1: number analyzed (Participants) | 34
  2 hours Post-Midday Dose, Week 1 | 35.00 (17.172)
  Pre-Morning Dose, Week 6: number analyzed (Participants) | 34
  Pre-Morning Dose, Week 6 | 19.99 (15.598)
  30 minutes Post-Morning Dose, Week 6: number analyzed (Participants) | 34
  30 minutes Post-Morning Dose, Week 6 | 24.50 (17.916)
  1 hour Post-Morning Dose, Week 6: number analyzed (Participants) | 34
  1 hour Post-Morning Dose, Week 6 | 24.68 (19.577)
  2 hours Post-Morning Dose, Week 6 | 26.79 (18.709)
  3 hours Post-Morning Dose, Week 6: number analyzed (Participants) | 34
  3 hours Post-Morning Dose, Week 6 | 26.40 (16.961)
  4 hours Post-Morning Dose, Week 6: number analyzed (Participants) | 34
  4 hours Post-Morning Dose, Week 6 | 24.04 (17.641)
  Pre-Midday Dose, Week 6: number analyzed (Participants) | 34
  Pre-Midday Dose, Week 6 | 17.15 (13.190)
  2 hours Post-Midday Dose, Week 6: number analyzed (Participants) | 34
  2 hours Post-Midday Dose, Week 6 | 25.49 (14.297)

17. Secondary Outcome: Pharmacokinetics: Ataluren Plasma Exposure in Ambulatory Participants
Description: Blood for ataluren concentrations were collected on Day 2 of Week 1 and Day 2 of Week 6. Analysis of the blood samples was to be conducted using a validated HPLC-MS/MS method with a LLOQ of 0.5 μg/mL. Plasma concentrations BQ is treated as 0 in the summary calculation.
Time Frame: as for outcome 16
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable plasma data. Participants who were ambulatory were able to walk ≥75 meters unassisted at screening.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 25
μg/mL
  Pre-Morning Dose, Week 1: number analyzed (Participants) | 24
  Pre-Morning Dose, Week 1 | 0 (0)
  30 minutes Post-Morning Dose, Week 1: number analyzed (Participants) | 24
  30 minutes Post-Morning Dose, Week 1 | 14.88 (10.771)
  1 hour Post-Morning Dose, Week 1: number analyzed (Participants) | 24
  1 hour Post-Morning Dose, Week 1 | 14.65 (9.608)
  2 hours Post-Morning Dose, Week 1: number analyzed (Participants) | 24
  2 hours Post-Morning Dose, Week 1 | 20.96 (12.648)
  3 hours Post-Dose, Week 1: number analyzed (Participants) | 24
  3 hours Post-Dose, Week 1 | 26.29 (15.853)
  4 hours Post-Morning Dose, Week 1: number analyzed (Participants) | 24
  4 hours Post-Morning Dose, Week 1 | 26.19 (14.531)
  Pre-Midday Dose, Week 1: number analyzed (Participants) | 24
  Pre-Midday Dose, Week 1 | 15.26 (10.238)
  2 hours Post-Midday Dose, Week 1: number analyzed (Participants) | 24
  2 hours Post-Midday Dose, Week 1 | 32.08 (17.977)
  Pre-Morning Dose, Week 6: number analyzed (Participants) | 24
  Pre-Morning Dose, Week 6 | 14.83 (10.032)
  30 minutes Post-Morning Dose, Week 6: number analyzed (Participants) | 24
  30 minutes Post-Morning Dose, Week 6 | 18.08 (8.654)
  1 hour Post-Morning Dose, Week 6: number analyzed (Participants) | 24
  1 hour Post-Morning Dose, Week 6 | 17.75 (8.660)
  2 hours Post-Morning Dose, Week 6: number analyzed (Participants) | 24
  2 hours Post-Morning Dose, Week 6 | 20.33 (9.103)
  3 hours Post-Morning Dose, Week 6: number analyzed (Participants) | 24
  3 hours Post-Morning Dose, Week 6 | 20.13 (9.423)
  4 hours Post-Morning Dose, Week 6: number analyzed (Participants) | 24
  4 hours Post-Morning Dose, Week 6 | 18.72 (12.255)
  Pre-Midday Dose, Week 6: number analyzed (Participants) | 24
  Pre-Midday Dose, Week 6 | 12.40 (6.775)
  2 hours Post-Midday Dose, Week 6: number analyzed (Participants) | 24
  2 hours Post-Midday Dose, Week 6 | 21.09 (7.959)

18. Secondary Outcome: Corticosteroid Plasma Concentrations as Assessed by a Validated Bioanalytical Method, in Participants Who Received a Daily Corticosteroid Regimen With Prednisone or Deflazacort
Description: Blood for prednisone and deflazacort concentrations were collected on Day 2 of Week 1 and Day 2 of Week 6. Plasma samples for the determination of prednisone concentrations were analyzed using a validated HPLC/MS/MS method, with LLOQs of 1.00 nanograms/milliliters (ng/mL). Prednisone concentrations <1.01 are treated as 1.01 in the summary calculation. Plasma samples for the determination of 21-desacetyl deflazacort concentrations were analyzed using a validated HPLC/MS/MS method with an LLOQ of 1.0 ng/mL. Deflazacort concentrations BQ are treated as 0 in the summary calculation.
Time Frame: as for outcome 16
Population: All enrolled participants who received at least 1 dose of study drug (As-Treated Population) and had evaluable prednisone or deflazacort plasma data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 36
ng/mL
  Pre-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  Pre-Dose, Prednisone, Week 1 | 1.01 (0)
  30 minutes Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  30 minutes Post-Dose, Prednisone, Week 1 | 18.27 (14.451)
  1 hour Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  1 hour Post-Dose, Prednisone, Week 1 | 35.48 (24.026)
  2 hours Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  2 hours Post-Dose, Prednisone, Week 1 | 32.41 (27.603)
  3 hours Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  3 hours Post-Dose, Prednisone, Week 1 | 57.12 (6.948)
  4 hours Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  4 hours Post-Dose, Prednisone, Week 1 | 49.44 (12.139)
  6 hours Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  6 hours Post-Dose, Prednisone, Week 1 | 31.41 (12.367)
  8 hours Post-Dose, Prednisone, Week 1: number analyzed (Participants) | 4
  8 hours Post-Dose, Prednisone, Week 1 | 15.59 (8.735)
  Pre-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  Pre-Dose, Prednisone, Week 6 | 1.01 (0)
  30 minutes Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  30 minutes Post-Dose, Prednisone, Week 6 | 17.13 (16.376)
  1 hour Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  1 hour Post-Dose, Prednisone, Week 6 | 32.48 (21.190)
  2 hours Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  2 hours Post-Dose, Prednisone, Week 6 | 39.91 (26.374)
  3 hours Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  3 hours Post-Dose, Prednisone, Week 6 | 41.02 (13.444)
  4 hours Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  4 hours Post-Dose, Prednisone, Week 6 | 38.82 (5.934)
  6 hours Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  6 hours Post-Dose, Prednisone, Week 6 | 24.95 (14.243)
  8 hours Post-Dose, Prednisone, Week 6: number analyzed (Participants) | 4
  8 hours Post-Dose, Prednisone, Week 6 | 13.52 (11.872)
  Pre-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  Pre-Dose, Deflazacort, Week 1 | 0 (0)
  30 minutes Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 19
  30 minutes Post-Dose, Deflazacort, Week 1 | 28.25 (31.968)
  1 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  1 hours Post-Dose, Deflazacort, Week 1 | 49.47 (43.631)
  2 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  2 hours Post-Dose, Deflazacort, Week 1 | 74.00 (49.349)
  3 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  3 hours Post-Dose, Deflazacort, Week 1 | 63.34 (38.045)
  4 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  4 hours Post-Dose, Deflazacort, Week 1 | 45.50 (31.427)
  6 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 20
  6 hours Post-Dose, Deflazacort, Week 1 | 18.67 (17.648)
  8 hours Post-Dose, Deflazacort, Week 1: number analyzed (Participants) | 19
  8 hours Post-Dose, Deflazacort, Week 1 | 7.57 (9.418)
  Pre-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  Pre-Dose, Deflazacort, Week 6 | 0.06 (0.268)
  30 minutes Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  30 minutes Post-Dose, Deflazacort, Week 6 | 33.46 (32.511)
  1 hour Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  1 hour Post-Dose, Deflazacort, Week 6 | 71.94 (77.370)
  2 hours Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  2 hours Post-Dose, Deflazacort, Week 6 | 81.41 (44.945)
  3 hours Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  3 hours Post-Dose, Deflazacort, Week 6 | 49.63 (26.633)
  4 hours Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  4 hours Post-Dose, Deflazacort, Week 6 | 25.85 (16.126)
  6 hours Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  6 hours Post-Dose, Deflazacort, Week 6 | 10.14 (14.080)
  8 hours Post-Dose, Deflazacort, Week 6: number analyzed (Participants) | 20
  8 hours Post-Dose, Deflazacort, Week 6 | 4.15 (7.985)

19. Secondary Outcome: Change in Muscle Composition as Assessed by Limb Magnetic Resonance (MR) Testing
Description: This Outcome Measure is an exploratory study objective and data were not collected or analyzed for this extension study.
Time Frame: Baseline, Week 48, Week 60
Population: All enrolled participants who received at least 1 dose of study drug and had Baseline and on-treatment data (Evaluable Population) with evaluable muscle composition data. Muscle composition data were not collected or analyzed for this extension study.
Arm/Group | Ataluren
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 89
Description: All enrolled participants who received at least 1 dose of study drug (As-Treated Population).
Arm/Group | Ataluren
Serious Adverse Events (participants affected / at risk) | 6/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren (N=36)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=36)
Myocardial fibrosis (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 3
Stomach discomfort (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 24
Asthenia (General disorders) | 3
Disease progression (General disorders) | 4
Gait disturbance (General disorders) | 4
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Influenza (Infections and infestations) | 5
Localized Infections (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 10
Contusion (Injury, poisoning and procedural complications) | 7
Excoriation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 11
Head injury (Injury, poisoning and procedural complications) | 3
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 5
Joint sprain (Injury, poisoning and procedural complications) | 5
Limb injury (Injury, poisoning and procedural complications) | 2
Postprocedural discomfort (Injury, poisoning and procedural complications) | 9
Procedural pain (Injury, poisoning and procedural complications) | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 2
Insulin resistance (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Scoliosis (Musculoskeletal and connective tissue disorders) | 5
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 17
Migraine (Nervous system disorders) | 4
Motor dysfunction (Nervous system disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 3
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the Sponsor for review. The Sponsor may consult with the PI to require changes to the communication or extend the embargo.